CLINICAL TRIAL: NCT06402253
Title: Social Media Artistic tRaining in Teenagers
Brief Title: A Music and Visual Arts Digital Intervention in Teenagers to Promote Healthy Engagement With Social Media.
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: American Composers Orchestra (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-FY2023-7419; 101063319 (Other Grant/Funding Number: European Research Council); 2023 (Other Grant/Funding Number: GRAMMY Museum Foundation)
Record Dates: First submitted 2024-04-15; First posted 2024-05-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Subjects; Mental Health Issue
Keywords: Mental health; Adolescents; Social media; Music; Neuroarts; Cognition; Brain imaging
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is organized around a 3-month digital music composition intervention for teenagers between 13 and 16 years old. This main music intervention will be compared with an active digital visual-art (i.e., photography) intervention, whose content is planned in parallel with the music one, and a passive no-intervention control group. The interventions will be administered in 24 sessions, with two 1-hour classes per week. Active interventions will cover both basic structural concepts (around music or photography, in each case) that will allow the participants to expand their understanding and appreciation of these kind of artistic stimuli; as well as hands-on experience in specific software for music / photography composition and edition (i.e., Soundtrap, Photoshop). Passive control participants will be monitored for 3-months and offered to complete one of the trainings after completing the study.
  All groups will complete evaluations before and after the 3-month interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Composition / Edition (Experimental): Teenage participants assigned to the 'Music Composition / Edition' (MUS) intervention will receive the 3-month Music Composition Intervention, completing self-reporting weekly measures of mood and social media usage, as well as a pre- and a post-intervention evaluation in which cognitive, mental-health, mood, social media usage and neuroimaging measures will be obtained.
  Interventions: Behavioral: Music composition / edition
- Photography Composition / Edition (Active Comparator): Teenage participants assigned to the 'Photography Composition / Edition' or Visual-Arts (VIS) intervention will receive the 3-month Photography Composition/Edition Intervention, completing self-reporting weekly measures of mood and social media usage, as well as a pre- and a post-intervention evaluation in which cognitive, mental-health, mood, social media usage and neuroimaging measures will be obtained.
  Interventions: Behavioral: Photography composition / edition
- Control (No Intervention): Teenage participants assigned to the 'Passive Control' (CON) arm will complete self-reporting weekly measures of mood and social media usage during 3 months, as well as a pre- and a post-intervention evaluation in which cognitive, mental-health, mood, social media usage and neuroimaging measures will be obtained.
  Once their participation in the study is complete, controls will be offered to complete the intervention of their choosing, according to the availability of teaching artists and locations to perform this.

INTERVENTIONS:
Behavioral: Music composition / edition — Participants in this group will complete two 1-hour music composition training intervention sessions per week over the course of 3 months (24 sessions total). These sessions will take place in the participating schools' premises, during normal hours corresponding to their advisory period class; or in participating centers during extracurricular activities' periods.
  The curriculum for these music composition lessons has been developed specifically for this project, in collaboration and based on the educational music composition programs from the American Composers Orchestra (ACO).
  Lessons review basic structural musical concepts, practicing active listening and music appreciation skills, teaching about the use of music-composition specific software (i.e., Soundtrap), and helping the students in expressing themselves / their identity through music, learning about musical story-telling through the creation of their own musical pieces from scratch.
  Other Names: MUS
  Arms: Music Composition / Edition
Behavioral: Photography composition / edition — Participants in this group will complete two 1-hour photography/visual-arts composition/edition intervention sessions per week over the course of 3 months (24 sessions total). These sessions will take place in the participating schools' premises, during normal hours corresponding to their advisory period class; or in participating centers during extracurricular activities' periods.
  The curriculum for these photography composition lessons has been developed specifically for this project, in collaboration and based on educational photography/film programs from Downtown Community TV Center (DCTV).
  Lessons review basic structural photography/visual-arts concepts, practicing visual-arts appreciation skills, teaching about the use of photography edition specific software (i.e., Photoshop), and helping the students in expressing themselves/their identity through photography, learning about visual story-telling through the creation of their own photographical projects from scratch.
  Other Names: VIS; Visual-arts Composition / Edition
  Arms: Photography Composition / Edition

SUMMARY:
The primary goal of this interventional study is to explore whether 3 months of arts-based digital interventions can change the way in which teenagers (13-16 years of age) use social media and are affected by them. The main questions it aims to answer are:

* Can we give teenagers new, stimulating, and more goal-oriented ways of using social media through arts-based digital trainings and active discussions around social media?
* Can these arts-based digital interventions also help teenagers to overcome the negative consequences of social media overuse (such as depression, anxiety, and reduced attention and cognitive performance)? Secondarily, this study also aims to explore the brain and behavioral traits associated with these arts-based interventions to better understand how they work.

Researchers will compare a music composition intervention with two other interventions: an active control intervention based on visual-arts instead of music (i.e., photography), and a passive approach to control for the mere pass of time.

Participants will:

* Complete a baseline and a post-intervention evaluation where researchers will obtain measures of cognitive performance (attention and executive functions, mainly), mood, mental health, brain structure and function, and social media usage and attitudes towards these platforms.
* Complete weekly measures regarding their use of social media platforms and their mood.
* Complete 3-month arts-based composition / edition intervention (based on music or visual-arts/photography), or the equivalent time with no intervention (passive control group).

The motivation of this study was driven by the observation that, in recent years, there has been an increasing use of social media and digital devices in teenagers, while the scientific community still does not fully understand the effects of the overuse of these digital means and platforms. Moreover, some of the negative effects described to be associated with the passive overuse of social media tap on the same brain structures that are benefited by musical and artistic trainings. Hence, we thought it could be worth trying to use arts-based training to help teenagers compensate for or overcome the negative effects of social media at the neural, cognitive, mood and mental health levels.

This study introduces novelty through three main aspects. Firstly, it employs a digital art creation approach that requires no classical art training, making it more accessible and less intimidating. Secondly, it incorporates commonly used digital devices (e.g., phones/tablets) and motivating environments into the learning process, integrating the development of new digital skills and the practice of critical thinking around the use of SM into normal classroom activities. Finally, the study employs a multi-methodological approach to explore the brain mechanisms underlying mental-health and cognitive changes resulting from arts-based interventions.

Finally, we believe that conclusions from SMART will:

* set the basis for developing preventive and therapeutic interventions for depression and anxiety in teenagers,
* promote educational programs that provide optimal tools for adolescents to navigate social media in a healthy manner, and
* inspire educational policy.

DETAILED DESCRIPTION:
1. Project Description Smart devices and social media (SM) have become prevalent among teenagers, raising questions about their effects on mental health and cognition. Most recent research has focused on the negative effects of SM overuse, including an increased risk of developing depression and anxiety, and alterations in cognitive functions, mainly attention. However, SM have also proven to have positive influences, such as promoting social interaction, creativity, and wellness, among others. Hence, the issue does not seem to be the time spent on SM per se, but the type of activity, content, and engagement the adolescents carry out on these platforms. As the U.S. Surgeon General recently warned, with the increasing use of smart devices and SM in youth, more resources must be dedicated to assessing which SM activities are beneficial or detrimental for the developing brain of adolescents.

   On the other hand, prior research suggests that art-based interventions, such as those based on music, improve mental health, and promote plastic changes in brain networks related to executive function and emotional regulation. Interestingly, these same brain areas and functions are known to be affected by SM passive overuse.

   Thus, here, the investigators use music and visual arts interventions to transform adolescent usage of SM, with the aim of mitigating the negative effects of excessive passive use of these platforms. The research team hypothesizes that both music and visual art interventions will improve mental health and enhance cognition. Further, researchers expect this cognitive and mental-health improvement to be paired with structural changes in brain centers related to emotional processing and executive function.
2. Research Question The main motivation and research question behind SMART is whether art appreciation and practice can change the way teenagers interact on SM, overcoming the negative influence of smart devices and social media platforms, and ultimately leading to beneficial cognitive and emotional effects. The first specific goal is to transform the use of social media in teenagers by providing them with digital (i.e., using software solutions) arts-based training, tools, and goal-oriented activities that they can implement in SM, while stimulating their critical thinking about these platforms. The investigators hypothesize that these tools and reflections will help the participants have a healthier relationship with SM, aiding them, for instance, to be critical about the content shared online, to look for healthier and more respectful online interactions, and/or to look for more stimulating activities to do online.

   The second specific goal would be to elucidate the behavioral and brain mechanisms behind the potential effects of music and visual-arts interventions on cognitive and emotional processing. Researchers expect the digital arts-based interventions to have positive effects on executive functions, specifically in the realm of attention, and on emotional and mental health markers. Investigators hypothesize that improvements in mental health will correlate with plastic changes in emotional and reward-related centers such as ventral striatum and ventromedial prefrontal cortex. Furthermore, the research team predicts that cognitive improvements will be related to plastic changes in prefrontal regions related to attention and executive functions.

   As secondary goals, SMART aims to develop art-related training programs that are useful, motivating, and applicable in educational contexts. Investigators would also like them to be applicable to preventive and therapeutic approaches aiming to improve the wellbeing and mental health of patients living with chronic conditions (such as diabetes, cancer, or major depression). Ultimately, the researchers aim to raise awareness of the benefits and importance that art-related activities, especially musical ones, have during development.
3. Research Applications Although some recent and currently ongoing investigations are also working on improving attention and executive functions in children and adolescents through cognitive training, even by using music and visual-arts interventions, the proposed project is the first of its kind in exploring the effects of arts-based training in transforming adolescents' use of SM. If predicted benefits from digital artistic interventions are confirmed, conclusions from SMART will have a ground-breaking impact in policy making regarding adolescents' mental health and education. Moreover, the conclusions and materials developed within this project have the potential to be applied in clinical contexts (e.g., health education, therapeutic purposes) in a wide array of physical and mental health conditions. For instance, arts-based interventions like the ones proposed here could be developed for the management of stress, depression, and anxiety symptoms associated with chronic health conditions such as diabetes or cancer.
4. Methodology High school students (9th graders; ages 13-16) will be recruited and divided into two intervention groups/arms: one focused on music composition/edition and another on photography composition/edition. An additional group that will not complete any intervention will be part of the study as a passive control. Participants will be recruited from Fort Hamilton High School (a public school in Brooklyn, NYC), and other public high schools in the NYC area with which collaboration agreements are being set nowadays. A pre-post longitudinal experimental design will be implemented. A sample size analysis determined that to have 80% of power to detect a large effect in a 2 (Pre/Post) x 3 (Group: Music, Visual Art, Control) mixed between-within repeated measures ANOVA, 18 participants per group are required. Investigators will recruit 30 participants per group to account for attrition. Individual experience in music and visual arts will be taken into account, mostly targeting non-experts but not excluding by that factor. Interventions will be administered in 1-hour sessions twice a week for 3 months (24 sessions; 3-month art-based interventions have been previously optimal at inducing mental health/cognitive improvements and brain plasticity. Interventions will include basic structural concepts from each discipline (musical, visual) so that participants are able to appreciate, edit, and create from scratch their own digital pieces, while maintaining a parallel structure and exigency between both types of interventions.

   Participants will create their artistic pieces using software such as SoundTrap/GarageBand (Music group) and LightRoom/Photoshop (Visual Art group). The classes will also include concepts related to the creative process, exploration of curiosity and identity within artistic activities, teamwork, and collaboration. SM will be used or included in discussions with the students every week to explore inspiration, reflect on what artists share online, be critical about how people comment online, and how to react to criticisms/feedback. The control group will not receive any musical or visual art training initially but will be able to complete the intervention of their choice once the study is over. The interventions will be taught by experienced instructors from the American Composers Orchestra (Music) and NYU's department of Integrated Design and Media (Visual Art).

   All participants will complete a baseline and a post-intervention 3-month follow-up evaluation that will include: (i) measures of mental health (via validated self-reports of depression, anxiety, general mood, and self-esteem); (ii) cognitive function (attention, measured via a flanker and a foraging inattentional blindness task); and (iii) brain plasticity, via the assessment of gray (GM) and white matter (WM) structure (MRI). Regarding the latter, researchers will collect high resolution T1-weighted images (1x1x1 mm3) for GM analysis and a diffusion-weighted MRI sequence for WM (1.5x1.5x1.5 mm3; 128 diffusion weighted volumes; b-value of 1500 s/mm2). The investigators will also collect information regarding participant's attitudes, opinions and usage of SM, and their sensitivity to general and artistic rewards. Continuous measures will include weekly input regarding: (i) progression of abilities and engagement in the arts classes (by instructors and main research, intervention groups); (ii) mood and motivation states (PANAS); and (iii) self-reported SM usage by filling the number of hours spent on their smartphones and the list and hours spent on their most-used apps (via their smartphone built-in screen-time function).

   Longitudinal changes in mental health and cognition will be assessed using JASP and a mixed within-between repeated measures 3x2 ANOVA. Post-hoc tests with Tukey correction for multiple comparisons will be used for significant main effects and interactions. Brain changes will be assessed via Voxel Based Morphometry as implemented in SPM12 and CAT12. FWE-correction will be used to control for multiple comparisons. For WM, researchers will use Tract-Based Spatial Statistics (TBSS) and will perform tractography of the main white matter pathways (e.g., arcuate, inferior longitudinal, uncinate, and inferior fronto-occipital fasciculi, corpus callosum, etc.) using Automatic Fiber Quantification. The investigators will assess markers of microstructural WM integrity previously related to cognitive and mental health status (Fractional Anisotropy, Axial, Radial, and Mean Diffusivity). FWE-correction using non-parametric permutations will be used to control for multiple comparisons. Spearman correlations will be used to assess the relationship between significant changes in mental health, cognitive, and brain plasticity.

   Regarding recruitment timelines, the researchers expect to have active groups recruited, completing the interventions during both the Fall 2024 and the Spring 2025 semesters, and take the Fall 2025 semester to work on finding matching controls and adjusting recruitment to compensate for the expected attrition rate of 20-30% of recruited participants.
5. Access and Dissemination Dissemination actions will target both the scientific community and the general public. All publications will be released as open access articles in international peer-reviewed scientific journals. All data and teaching materials from both interventions will be released as open-access resources. Also, to raise awareness about the issues that could be improved by exploiting SMART results, white papers directed to education/culture policy makers will also be published. Oral and poster presentations at renowned international conferences, such as Human Brain Mapping and Society for Neuroscience, are also planned. Actually, this protocol has been accepted to be presented as a poster at the "Music and Neuroscience VIII" conference that will be held in Helsinki in June 2024 (this is the most important event for the neuroscience of music research, held every 3 years).

Also, SMART 1-day workshops at local schools will be held targeting parents, teachers and educators, as well as policy makers. These workshops will explain the rationale and the project characteristics and results obtained up to that moment and will be used to hold open discussions with attendants to solve doubts and fully understand stakeholders' interests and concerns. These discussions could also motivate future work and an expansion of the current intervention protocol/study. The research team is currently working on the setup of the SMART website and Social Media accounts, aiming to inform and keep up to date both the scientific community and the general population regarding the development of the project. Finally, participation on national and international science outreach activities, such as science fairs and conferences at public and private schools and science popularization articles published in online dedicated platforms (i.e., The Conversation, Naukas), are ensured thanks to the ongoing involvement of Dr. Vaquero in these types of activities.

ELIGIBILITY:
INCLUSION CRITERIA:

* We are not concerned with country of birth, native language, race, or gender. Furthermore, we will not exclude subjects based on their neurodevelopmental, neurological, or psychiatric disorders, or based on their background or previous training in music, visual/plastic arts, or film/multimedia.
* We will recruit participants who are 13-16 years old.
* If they agree to participate in the neuroimaging sessions, participants will not have any contraindications for completing MEG or MRI scans.
* In addition, we intend to recruit the parents of child participants to answer questions about their child. For these participants, we have no inclusion criteria except that they are the parent of a child participating in the study.

EXCLUSION CRITERIA:

* We will exclude participants who are not between the ages of 13 and 16 years old.
* For the additional neuroimaging measures, we will exclude participants who have any contraindications for MEG or MRI if they choose to participate in the optional MEG and MRI scans.
* For recruiting parents, we will exclude those who are not parents of a child enrolled in the study.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Post - Pre changes in attitudes and importance given to social media | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  qualitative differences in attitudes and importance of SM self-reported by participants before and after the intervention. Researchers will use a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire').
Post - Pre changes in social media profiles followed in social media | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  qualitative differences in the kind of profiles followed by participants before and after the intervention. Researchers will use a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire').
Post - Pre changes in mood and emotional reaction while being online | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  qualitative differences in participants' mood and emotional reaction while using social media before and after the intervention. Researchers will use a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire').
Weekly evolution of screentime | From week 1 to week 12 of the intervention (or 3-month no intervention period for the control group).
  measures of actual smartphone usage will be collected every week during the intervention period (or the 3-month period, in the case of the passive Control group) via self-report questionnaires in which participants will fill the objective smartphone screentime usage data measured by the screentime function on their device. The higher the value input here by participants, the greater the amount of hours spent on their phone.
Weekly evolution of mood | From week 1 to week 12 of the intervention (or 3-month no intervention period for the control group).
  measures of weekly mood will be gathered by making participants fill the Positive and Negative Affect Scale (PANAS) once a week. This scale ranges from 10 to 50 for Positive Affect, with greater values meaning greater presence of positive mood; and from 10 to 50 for Negative Affect, with greater values meaning greater presence of negative mood.
Post - Pre changes in self-esteem | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  the investigators will use the standard test Rosenberg Self-Esteem Questionnaire, ranging from 0 to 30, with scores between 15 and 25 pertaining to a normal range and scores below 15 suggesting low self-esteem.
Post - Pre changes in Depression (CDI) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the Children Depression Inventory (CDI), a 27-item scale ranging from 0 to 54. The higher the CDI score, the higher the depressive state.
Post - Pre changes in Anxiety (SCARED) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the Screen for Child Anxiety Related Disorders (SCARED), a scale ranging from 0 to 82 with values greater than 25 in the total score indicating the presence of anxiety disorder. It is divided in subscales for Panic Disorder (cut-off=7), Generalized Anxiety Disorder (cut-off=9), Separation Anxiety Disorder (cut-off=5), Social Anxiety Disorder (cut-off=8), and School Avoidance (cut-off=3).
Post - Pre changes in Mood | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measures of mood will be acquired by using the Positive and Negative Affective Scale (PANAS). This scale ranges from 10 to 50 for Positive Affect, with greater values meaning greater presence of positive mood; and from 10 to 50 for Negative Affect, with greater values meaning greater presence of negative mood.
Post - Pre changes in Attention | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via an Attentional Flanker task, a specifically developed task for this purpose measuring accuracy and reaction times for congruent, incongruent, and neutral trials.
Post - Pre changes in verbal learning and memory | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  researchers will apply the Rey's Auditory Verbal Learning test (AVLT), a standard test counting number of remembered words in each immediate trial and after a delay of 20 minutes. The higher the number in each trial, the better the participant's verbal and learning functions
Post - Pre changes in auditory working memory | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the WAIS-V Letter Number Sequencing. Score ranges from 0 to 21, with higher scores indicating better auditory working memory.
Post - Pre changes in functional connectivity at rest | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured using functional MRI (fMRI). Summary beta values representing the level of brain activity will be calculated in functional networks of interest.
Post - Pre changes in neurophysiological correlates of pre-attentive auditory detection | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  the Mismatch Negativity (MMN) component would be characterized for each melodic and rhythmic violation of the presented stimuli. The amplitude of the MMN would be calculated and compared between timepoints.
Post - Pre changes in brain morphology / anatomy | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  Using structural Magnetic Resonance Imaging, researchers will obtain T1-weighted images that will allow for the study of participants' cortical and subcortical gray matter. Applying analyses such as Voxel-Based Morphometry or Cortical Thickness values of gray matter will be obtained, compared between groups and correlated with other types of measures (i.e., cognitive, mental health, behavioral).
Post - Pre changes in brain structural connectivity | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  Using structural Magnetic Resonance Imaging, researchers will obtain diffusion-weighted images that will allow for the study of participants' white matter structural connectivity between areas of interest. Applying analyses such Tract-Based Spatial Statistics or Tractographical reconstruction of white-matter pathways, macro- and microstructural measures of tracts of interest will be calculated, compared between groups and correlated with other types of measures (i.e., cognitive, mental health, behavioral).

SECONDARY OUTCOMES:
Treatment Fidelity | From beginning of the intervention to end of intervention (at week 12)
  Treatment fidelity will be annotated for every week and session as a percentage that represents the accuracy and fit between the actual lessons carried out and the original planned lesson for each intervention session. This percentage will be estimated by the research team present at each intervention session.
Students' Engagement during Interventions | From beginning of the intervention to end of intervention (at week 12)
  Attendance and engagement during every lesson will be recorded and valued using a 1-7 Likert scale. These observations and ratings will be annotated by the research team present at each intervention session.
Post - Pre changes in self-reported screentime | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  the investigators will use a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire'). The higher the value input here by participants, the greater the amount of hours spent on their phone.
Post - Pre changes in social media platforms used | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  qualitative change in students' top 10 self-reported most-used apps in a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire').
Post - Pre changes in types of posts shared online | From enrollment to the end of the post-intervention evaluation (roughly at week 14).
  qualitative differences in the types of posts shared by participants in the social media profiles before and after the intervention. Researchers will use a questionnaire specifically developed for this purpose ('Usage, Attitudes & Opinions about Social Media Questionnaire').
Weekly evolution of apps most used during weekday | From week 1 to week 12 of the intervention (or 3-month no intervention period for the control group).
  measures of actual most-used apps during a given weekday will be collected every week during the intervention period (or the 3-month period, in the case of the passive Control group) via self-report questionnaires in which participants will fill the objective list of most-used app days during the given weekday and for how long has each of them been used, measured by the screentime function on participants' device.
Weekly evolution of apps most used during weekend day | From week 1 to week 12 of the intervention (or 3-month no intervention period for the control group).
  measures of actual most-used apps during a given weekend day will be collected every week during the intervention period (or the 3-month period, in the case of the passive Control group) via self-report questionnaires in which participants will fill the objective list of most-used app days during the given weekend day and for how long has each of them been used, measured by the screentime function on participants' device.
Post - Pre changes in Depression (DASS21) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the Depression, Anxiety and Stress Scale 21 (DASS-21), with 7 items dedicated to measure Depression. Scores range from 0 to 42, with higher scores indicating greater depressive symptoms (scores 14-20 suggest moderate depression, scores greater than 28 suggest extremely severe depression)
Post - Pre changes in Anxiety (DASS21) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the Depression, Anxiety and Stress Scale 21 (DASS-21), with 7 items dedicated to measure Anxiety. Scores range from 0 to 42, with higher scores indicating greater anxiety symptoms (scores 10-14 suggest moderate anxiety, scores greater than 20 suggest extremely severe anxiety).
Post - Pre changes in Stress (DASS21) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured via the Depression, Anxiety and Stress Scale 21 (DASS-21), with 7 items dedicated to measure Stress. Scores range from 0 to 42, with higher scores indicating greater stress symptoms (scores 19-25 suggest moderate stress, scores greater than 34 suggest extremely severe stress).
Post - Pre changes in the Total Mood Disturbance (POMS) | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  researchers will use the Profile of Mood and States Scale (POMS) with a total mood disturbance measure calculated out of summing up the negative-mood subscales (Anger-Hostility: 0- 20; Confusion-Bewilderment: 0 - 20; Depression-Dejection: 0 - 28; Fatigue-Inertia: 0 - 20; Tension-Anxiety: 0 - 24) and subtract the positive mood subscale (Vigor-Activity: 0 - 24). The higher the scores the greater the probability of having a mood-related issue.
Post - Pre changes in Social Anxiety | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  researchers will use the Social Anxiety Scale for Adolescents (SAS-A), a 18-item scale whose scores range from 18 to 90 in the total SAS-A score (but that also counts with subscales in Fear of Negative Evaluation: 8-40; Social Avoidance and Distress - New: 6-30; and Social Avoidance and Distress - General: 4-20). The higher the scores, the greater the social anxiety symptoms (recommended cut-off=50).
Post - Pre changes in Focused Attention and Executive Functions | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  researchers have specifically developed the Foraging Inattentional Blindness task for this purpose. Visual targets and distractors move around the screen, and participants have to find the targets as quickly as possible until reaching a total score of 200 points. Reaction times and search strategy within the screen are recorded.
Post - Pre changes in functional connectivity at rest within different frequency bands | Difference from enrollment to the end of the post-intervention evaluation (roughly at week 14).
  measured using Magnetoencephalography (MEG), connectivity at rest between brain sources of interest will be calculated within different frequency bands.

OTHER OUTCOMES:
Students' Feedback about the Intervention | End of intervention (week 12)
  At the end of the intervention, students will have to fill a questionnaire in order to rate their likeness and express their opinions about the intervention program in which they have participated. We will use a questionnaire specifically developed for this purpose.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fort Hamilton High School, Brooklyn, New York
  - Faculty of Arts & Science, Psychology Department - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU. Requests may be directed to: pripolles@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Study Protocol Intervention Program Curriculum Statistical Analysis Plan (SAP) Anonymized Behavioral and Neuroimaging Data Metadata / Workflows Pre-prints
URL: https://datadryad.org/

REFERENCES:
- [Background] Ripolles P, Rojo N, Grau-Sanchez J, Amengual JL, Camara E, Marco-Pallares J, Juncadella M, Vaquero L, Rubio F, Duarte E, Garrido C, Altenmuller E, Munte TF, Rodriguez-Fornells A. Music supported therapy promotes motor plasticity in individuals with chronic stroke. Brain Imaging Behav. 2016 Dec;10(4):1289-1307. doi: 10.1007/s11682-015-9498-x. PMID 26707190
- [Background] Siponkoski ST, Martinez-Molina N, Kuusela L, Laitinen S, Holma M, Ahlfors M, Jordan-Kilkki P, Ala-Kauhaluoma K, Melkas S, Pekkola J, Rodriguez-Fornells A, Laine M, Ylinen A, Rantanen P, Koskinen S, Lipsanen J, Sarkamo T. Music Therapy Enhances Executive Functions and Prefrontal Structural Neuroplasticity after Traumatic Brain Injury: Evidence from a Randomized Controlled Trial. J Neurotrauma. 2020 Feb 15;37(4):618-634. doi: 10.1089/neu.2019.6413. Epub 2019 Dec 5. PMID 31642408
- [Background] Bianco V, Berchicci M, Gigante E, Perri RL, Quinzi F, Mussini E, Di Russo F. Brain Plasticity Induced by Musical Expertise on Proactive and Reactive Cognitive Functions. Neuroscience. 2022 Feb 10;483:1-12. doi: 10.1016/j.neuroscience.2021.12.032. Epub 2021 Dec 29. PMID 34973386
- [Background] Vaquero L, Rodriguez-Fornells A, Reiterer SM. The Left, The Better: White-Matter Brain Integrity Predicts Foreign Language Imitation Ability. Cereb Cortex. 2017 Aug 1;27(8):3906-3917. doi: 10.1093/cercor/bhw199. PMID 27461123
- [Background] Simo M, Vaquero L, Ripolles P, Gurtubay-Antolin A, Jove J, Navarro A, Cardenal F, Bruna J, Rodriguez-Fornells A. Longitudinal Brain Changes Associated with Prophylactic Cranial Irradiation in Lung Cancer. J Thorac Oncol. 2016 Apr;11(4):475-86. doi: 10.1016/j.jtho.2015.12.110. Epub 2016 Jan 22. PMID 26804637
- [Background] Vaquero L, Rodriguez-Fornells A, Pera-Jambrina MA, Bruna J, Simo M. Plasticity in bilateral hippocampi after a 3-month physical activity programme in lung cancer patients. Eur J Neurol. 2021 Apr;28(4):1324-1333. doi: 10.1111/ene.14670. Epub 2020 Dec 30. PMID 33296534
- [Background] Vaquero L, Hartmann K, Ripolles P, Rojo N, Sierpowska J, Francois C, Camara E, van Vugt FT, Mohammadi B, Samii A, Munte TF, Rodriguez-Fornells A, Altenmuller E. Structural neuroplasticity in expert pianists depends on the age of musical training onset. Neuroimage. 2016 Feb 1;126:106-19. doi: 10.1016/j.neuroimage.2015.11.008. Epub 2015 Nov 14. PMID 26584868
- [Background] Gil-Gomez de Liano B, Quiros-Godoy M, Perez-Hernandez E, Wolfe JM. Efficiency and accuracy of visual search develop at different rates from early childhood through early adulthood. Psychon Bull Rev. 2020 Jun;27(3):504-511. doi: 10.3758/s13423-020-01712-z. PMID 32043221
- [Background] Mas-Herrero E, Singer N, Ferreri L, McPhee M, Zatorre RJ, Ripolles P. Music engagement is negatively correlated with depressive symptoms during the COVID-19 pandemic via reward-related mechanisms. Ann N Y Acad Sci. 2023 Jan;1519(1):186-198. doi: 10.1111/nyas.14931. Epub 2022 Nov 19. PMID 36401802
- [Background] Lu J, Moussard A, Guo S, Lee Y, Bidelman GM, Moreno S, Skrotzki C, Bugos J, Shen D, Yao D, Alain C. Music training modulates theta brain oscillations associated with response suppression. Ann N Y Acad Sci. 2022 Oct;1516(1):212-221. doi: 10.1111/nyas.14861. Epub 2022 Jul 19. PMID 35854670
- [Background] James CE, Tingaud M, Laera G, Guedj C, Zuber S, Diambrini Palazzi R, Vukovic S, Richiardi J, Kliegel M, Marie D. Cognitive enrichment through art: a randomized controlled trial on the effect of music or visual arts group practice on cognitive and brain development of young children. BMC Complement Med Ther. 2024 Apr 4;24(1):141. doi: 10.1186/s12906-024-04433-1. PMID 38575952
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Background] Orpella J., Bowling D., Tomaino C., Ripolles P. (2023). Effects of Affectively Parameterized Music on Mood and Attention. PsyArXiv. https://doi.org/10.31234/osf.io/yauxt.
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Sihvonen AJ, Leo V, Ripolles P, Lehtovaara T, Ylonen A, Rajanaro P, Laitinen S, Forsblom A, Saunavaara J, Autti T, Laine M, Rodriguez-Fornells A, Tervaniemi M, Soinila S, Sarkamo T. Vocal music enhances memory and language recovery after stroke: pooled results from two RCTs. Ann Clin Transl Neurol. 2020 Nov;7(11):2272-2287. doi: 10.1002/acn3.51217. Epub 2020 Oct 6. PMID 33022148
- [Background] Sarkamo T, Ripolles P, Vepsalainen H, Autti T, Silvennoinen HM, Salli E, Laitinen S, Forsblom A, Soinila S, Rodriguez-Fornells A. Structural changes induced by daily music listening in the recovering brain after middle cerebral artery stroke: a voxel-based morphometry study. Front Hum Neurosci. 2014 Apr 17;8:245. doi: 10.3389/fnhum.2014.00245. eCollection 2014. PMID 24860466
- [Background] Smout A, Chapman C, Mather M, Slade T, Teesson M, Newton N. It's the Content That Counts: Longitudinal Associations between Social Media Use, Parental Monitoring, and Alcohol Use in an Australian Sample of Adolescents Aged 13 to 16 Years. Int J Environ Res Public Health. 2021 Jul 16;18(14):7599. doi: 10.3390/ijerph18147599. PMID 34300049
- [Background] K Kaye L, Orben A, A Ellis D, C Hunter S, Houghton S. The Conceptual and Methodological Mayhem of "Screen Time". Int J Environ Res Public Health. 2020 May 22;17(10):3661. doi: 10.3390/ijerph17103661. PMID 32456054
- [Background] O'Reilly M, Dogra N, Hughes J, Reilly P, George R, Whiteman N. Potential of social media in promoting mental health in adolescents. Health Promot Int. 2019 Oct 1;34(5):981-991. doi: 10.1093/heapro/day056. PMID 30060043
- [Background] Mahalingham T, Howell J, Clarke PJF. Attention control moderates the relationship between social media use and psychological distress. J Affect Disord. 2022 Jan 15;297:536-541. doi: 10.1016/j.jad.2021.10.071. Epub 2021 Oct 26. PMID 34715177
- [Background] Wacks Y, Weinstein AM. Excessive Smartphone Use Is Associated With Health Problems in Adolescents and Young Adults. Front Psychiatry. 2021 May 28;12:669042. doi: 10.3389/fpsyt.2021.669042. eCollection 2021. PMID 34140904
- [Background] Camunas N, Mavrou I, Vaillo M, Martinez RM. An executive function training programme to promote behavioural and emotional control of children and adolescents in foster care in Spain. Trends Neurosci Educ. 2022 Jun;27:100175. doi: 10.1016/j.tine.2022.100175. Epub 2022 Mar 20. PMID 35501027
- [Derived] Vaquero L, Groves K, Munoz-Vidal EL, James K, Marlor JL, McIntyre C, Ostia L, Sirota S, Shields L, Dege F, Garcia-Mingo E, Ripolles P. Studying the effects of digital arts-based interventions on teenagers' social media usage, brain connectivity, and mental health: study protocol of the SMART project. Eur J Psychotraumatol. 2025 Dec;16(1):2550079. doi: 10.1080/20008066.2025.2550079. Epub 2025 Sep 17. PMID 40958721